CLINICAL TRIAL: NCT03272178
Title: Impact of Component Design and Fixation in Bone Remodeling After Total Knee Arthroplasty
Brief Title: Impact of Component Design and Fixation in Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor
Other Study IDs: 201708094
Record Dates: First submitted 2017-08-22; First posted 2017-09-05 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Arthroplasties, Knee Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Triathlon knee total knee arthroplasty: 50 Patients who are assigned to Triathlon knee, half cemented/half cementless
  Interventions: Device: Triathlon total knee implant
- Depuy knee total knee arthroplasty: 50 Patients who are assigned to Depuy knee, half cemented/half cementless
  Interventions: Device: Depuy total knee implant

INTERVENTIONS:
Device: Depuy total knee implant — patients from Dr Nunley's clinic will get a Depuy implant
  Groups: Depuy knee total knee arthroplasty
Device: Triathlon total knee implant — patients from Dr Barrack's clinic will get a Triathlon implant
  Groups: Triathlon knee total knee arthroplasty

SUMMARY:
The purpose of this study is to determine implant design and determine if method of fixation cemented versus cementless results in different bone loss patterns. The investigators also want to determine if clinical outcomes correlate with bone density changes.

DETAILED DESCRIPTION:
Patients who present to the clinical practices of Dr. Ryan Nunley and Dr. Robert Barrack and are suitable candidates for primary total knee arthroplasty(TKA) type assigned either cemented or cementless and Triathlon knee or Depuy by surgeon will be screened for eligibility and invited to participate. Data collected for the study will include standard of care clinical and radiographic evaluations collected during office visits and surgery, Dual Energy X-Ray Absorptiometry(DEXA) Bone density monitoring, as well as study-specific patient questionnaires. Clinical, radiographic and questionnaire data will be collected pre-operatively, at the time of surgery, and at 6 weeks, 1 year and beyond, and 2 years and beyond post-operatively. Patients will complete the following outcomes questionnaires preoperatively: New Knee Society Score, Oxford Knee Score, UCLA Activity Score, SF-12, and EQ-5D. The following questionnaires will be collected at four to six weeks, six months, one year and beyond, and two years and beyond postoperatively: New Knee Society Score, Forgotten Joint Score, Washington University Knee Satisfaction and Function Questionnaire, Oxford Knee Score, UCLA Activity Score, SF-12, and EQ-5D, and a Pain Drawing.

ELIGIBILITY:
Inclusion Criteria:

* Patients who qualify for a Primary Total knee using Triathlon Implant(thin tray) or Depuy Attune(thick tray) Implant
* 18-75 years of age
* Willing to sign informed consent
* Willing to return for all follow-up visits

Exclusion Criteria:

* Patients with inflammatory arthritis
* BMI > 40
* Patient with an active infection or suspected infection in the joint
* Patient who have undergone osteotomy
* Patients who have a previous diagnosis of osteopenia/osteoporosis or patients with weak bones and/or currently on medications to increase bone density/who have poor bone quality
* Patients who have had previous patella fracture or surgery
* Patients who have had previous knee or hip replacement surgery on the ipsilateral side
* Patients who require patellar resurfacing
* Patient with major medical/muscular/orthopedic deformities
* Unable to undergo DEXA scanning.
* Female patients of childbearing potential and an interest in getting pregnant in the future *NOTE: Patients receiving simultaneous bilateral total knee arthroplasties are eligible. Both knees are eligible for enrollment as long as all other inclusion/exclusion criteria are met for each knee. If only one knee is eligible it will be included. Patients receiving staged bilaterals are also eligible, provided that each knee meets the inclusion exclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A. Patients who qualify for a Primary Total Knee Arthroplasty using Stryker Triathlon Implant(thin tray) or Depuy Attune(thick tray) Implant
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Change in bone density | 2 years
  Patients will have a DEXA scan to look for change in bone loss at 6 weeks, 1 year, and 2 year to determine bone loss patterns and geometry

SECONDARY OUTCOMES:
knee society score | 2 years
  Knee society score questionnaire will be completed preoperatively, 6 weeks, 1 year, and 2 year.
Forgotten joint score | 2 years
  Forgotten join score questionnaire will be completed preoperatively, 6 weeks, 1 year, and 2 year.
Oxford knee score | 2 years
  Oxford knee score questionnaire will be completed preoperatively, 6 weeks, 1 year, and 2 year.
UCLA Activity score | 2 years
  UCLA questionnaire will be completed preoperatively, 6 weeks, 1 year, and 2 year.
SF-12 | 2 years
  SF-12 questionnaire will be completed preoperatively, 6 weeks, 1 year, and 2 year.
EQ-5D | 2 years
  EQ-5D questionnaire will be completed preoperatively, 6 weeks, 1 year, and 2 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States